CLINICAL TRIAL: NCT01549301
Title: Evaluation of Pharmacokinetic and Pharmacodynamic Parameters of Filgrastim (G-CSF)Produced by Blausiegel Indústria e Comércio Ltda. Compared to Granulokine Produced by Produtos Roche Químicos e Farmacêuticos S/A.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FILBLA1211I; Version 01 - 09/12/2011
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Filgrastim

ARMS (4):
- Group D 10 i.v. (Experimental): Two periods, crossover, single dose, i.v., 10 mcg, Comparator (n=16) x Test (n=16) in the first period and Test (n=16) x Comparator (n=16) in the second period, in a crossover basis.
  Interventions: Drug: Filgrastim
- Group C 5 i.v. (Experimental): Two periods, crossover, single dose, i.v., 5 mcg, Comparator (n=16) x Test (n=16) in the first period and Test (n=16) x Comparator (n=16) in the second period, in a crossover basis.
  Interventions: Drug: Filgrastim
- Group B 10 s.c. (Experimental): Two periods, crossover, single dose, s.c., 10 mcg/kg, Comparator (n=16) x Test (n=16) in the first period and Test (n=16) x Comparator (n=16) in the second period, in a crossover basis.
  Interventions: Drug: Filgrastim
- Group A 5 s.c. (Experimental): Two periods, crossover, single dose, s.c., 5 mcg, Comparator (n=16) x Test (n=16) in the first period and Test (n=16) x Comparator (n=16) in the second period, in a crossover basis.
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Filgrastim — filgrastim, single dose, s.c., dosage: 5 mcg/kg
  Arms: Group A 5 s.c.
Drug: Filgrastim — filgrastim, single dose, s.c., dosage: 10 mcg/kg
  Arms: Group B 10 s.c.
Drug: Filgrastim — Filgrastim, i.v., single dose, dosage: 5 mcg/kg
  Arms: Group C 5 i.v.
Drug: Filgrastim — Filgrastim, i.v., single dose, dosage: 10 mcg/kg
  Arms: Group D 10 i.v.

SUMMARY:
The primary aim of this study is to compare the pharmacokinetic and pharmacodynamic effects of two commercial preparations of filgrastim (T and C), after single dose via subcutaneous or intravenous administration at a concentration of 5 mcg/kg or 10 mcg/kg in healthy subjects through the alteration in the pharmacokinetic and pharmacodynamic parameters (measurement of serum levels of G-CSF and absolute neutrophil count - ANC).

ELIGIBILITY:
Inclusion Criteria:

* Agree with all study procedures, sign and date back by their own free will, the IC;
* Be between 18 and 50 years, of both sexes;
* Present a body mass index (BMI) greater than or equal to 20 and less than or equal to 28;
* are considered healthy, clinical, psychological and laboratory;
* are female, but they have and maintain a safe method of contraception during the study.

Exclusion Criteria:

* Known hypersensitivity to filgrastim;
* Hypersensitivity to products derived from E. coli;
* fever or infectious disease in the 07 days preceding the first administration;
* Positive serology for hepatitis B or C and HIV;
* Prior treatment with CSFs, interleukins and interferons;
* Participation in a clinical study in the last 12 months;
* Donation or loss of blood in the 03 months preceding the study;
* General anesthesia in the 03 months preceding the study;
* Provide a history of alcohol abuse, drug or drugs;
* Have a history of liver disease, renal, pulmonary, gastrointestinal, hematological, psoriasis, gout, acute myocardial infarction, thyroid or psychiatric disease;
* Pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameters will be based on the investigation of pharmacokinetics and pharmacodynamics of filgrastim in research subjects after administration of single dose via sc or iv routes at doses of 5 or 10 mcg/kg of the drug. | • PK.: 0, 15 min., 30 min., 45 min., 1h, 1h e 30min., 2h, 3h, 4h, 6h, 8h,10h, 12h, 16h, 24h and 48h. • PD (ANC): 0, 30 min., 1h, 2h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 32h, 48h, 72h, 96h and 120h

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil